CLINICAL TRIAL: NCT01322399
Title: Structural Integration for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Lab, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-000014; SRH; K01AT004916 (NIH)
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Back Pain Lower Back Chronic
Keywords: low back pain; chronic pain; manual therapy; Structural Integration
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Musculoskeletal Manipulations; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structural Integration plus usual care (Experimental): Each subject in this arm will receive ten Structural Integration treatments at intervals of between one and three weeks, and will also receive usual care for chronic low back pain as standard practice at Spaulding Medford Rehabilitation Clinic, which may include pain medication, exercise and physical therapy. Usual care will be provided on average twice weekly for between 3 and 7 weeks, at the discretion of the clinic's medical director
  Interventions: Procedure: Structural Integration; Procedure: Usual care
- Usual care (Active Comparator): Each subject in this arm will receive care for chronic low back pain as standard practice at Spaulding Medford Rehabilitation Clinic, which may include pain medication, exercise and physical therapy. Usual care will be provided on average twice weekly for between 3 and 7 weeks, at the discretion of the clinic's medical director
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Structural Integration — Structural Integration (SI) is an alternative method of manual therapy and somato-sensory training that purports to improve biomechanical functioning of the body as a whole rather than to focus on the treatment of specific symptoms. SI therapists employ both manipulation and somatosensory education. SI is delivered in a series of ten treatments, referred to as "the Ten Series," each of approximately one hour in duration. The Ten Series protocol includes manipulation of all major joints and anatomical segments. Each of the ten sessions aims to achieve a different set of biomechanical changes, which are regarded as contributing to the progressive approximation of specific ideals of posture and movement.
  Other Names: Rolfing, a registered service mark of the Rolf Institute
  Arms: Structural Integration plus usual care
Procedure: Usual care — Usual care in this study consists of the treatment regimen provided for chronic low back pain at Spaulding Medford Rehabilitation clinic, which may include pain medication, exercise and physical therapy. Frequency of treatment averages twice weekly, duration ranges from 3 to 7 weeks
  Other Names: Standard care

SUMMARY:
The primary purpose of study is the collection of feasibility data for a larger trial of Structural Integration (SI)(an alternative manual therapy) for chronic low back pain. The secondary purpose is the collection of preliminary data on 1) the therapeutic effect of SI plus usual care versus usual care alone - the hypothesis being the the effect size will be significantly greater in the SI plus usual care arm; and on 2) specific hypothesized mechanisms of that hypothesized therapeutic effect: a) improvements in cognitive behavioral factors; b) improvements in standing balance and gait, and c) improvements in selected blood biomarkers.

DETAILED DESCRIPTION:
Chronic, non-specific low back pain is among the most burdensome health problems in both prevalence and cost of care. Up to one third of acute low back pain cases may become chronic and lead to disability. A large fraction of chronic cases are absent of findings of well-understood causes, i.e. neoplastic, infectious or inflammatory conditions, or nerve compression, and are generally designated as "uncomplicated," "non-specific," or "mechanical." Usual care typically includes oral and injected medication, physical therapy and exercise. Therapeutic response is difficult to predict and many outcomes are unsatisfactory, with high rates of relapse.

Structural Integration (SI) is an alternative method of manual therapy and somato-sensory training that purports to improve the biomechanical functioning of the body as a whole rather than to focus on the treatment of specific symptoms. SI is delivered in a series of ten treatments, referred to as "the Ten Series," each of approximately one hour in duration. The Ten Series protocol includes manipulation of all major joints and anatomical segments. Each of the ten sessions aims to achieve a different, specified set of biomechanical changes which are regarded as contributing to the progressive approximation of specific ideals of posture and movement.

Forty (40) subjects will be recruited from among individuals entering treatment for chronic low back pain at outpatient rehabilitation clinics in the Boston area. Following baseline measures, subjects will be randomized with equal probability (50/50) to usual care alone versus usual care plus ten sessions of SI. SI treatment will be provided by qualified SI therapists at their private practice offices. They will be supervised on a monthly basis by a co-investigator with extensive prior experience in the clinical practice of SI.

Data will be collected at baseline, end-of-treatment, and endpoint. Baseline data will be collected prior to the subject's first treatment appointment, and endpoint data will be collected from all subjects at 20 weeks post-baseline. End-of-treatment measures will be conducted during the week following each subject's completion of their assigned treatment arm. Consequently, the average time elapsed between baseline and end-of-treatment will differ across the two treatment arms, because of different amounts of time allowed for the completion of usual care alone (3-7 weeks) versus usual care plus SI (10-15) weeks.

Analysis relevant to the primary aim of the study will be conducted as follows: The demographic characteristics of candidates referred, subjects enrolled, and dropouts will described. Descriptive statistics, both aggregate and per treatment arm, will be computed for data on retention and compliance with treatment, and on the use of concurrent medications. Each adverse events will be characterized by subject demographics and by treatment arm, and will also be rated for severity, likelihood of relation to the study, and expected versus unexpected.

Analysis relevant to the secondary aim of the study will be conducted as follows: Baseline to endpoint changes in therapeutic outcomes, cognitive-behavioral measures and blood assay values will be compared across treatment arms using appropriate statistical tests. Baseline to endpoint changes in standing balance and gait parameters will be analyzed using methods that are standard in the current literature. In addition to appropriate statistical tests, these include the visual inspection of graphic displays of the phase relationships between rotational movements of body segments during gait. The association between each mechanistic parameter - cognitive-behavioral, biomechanical, and blood biomarkers - and the primary and secondary therapeutic outcomes will be explored per treatment arm and in aggregate.

Data on changes between baseline and end-of-treatment will be subject to exploratory analysis within treatment arms only. Comparison across arms is inappropriate because of systematic variation in the average duration of treatment in usual care alone (estimated at 5 weeks) versus usual care plus SI (estimated at 12.5 weeks). Analysis will include the exploration of associations between changes in therapeutic outcomes on one hand, and mechanistic parameters on the other, but only within each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain patient-rated >=3 on a VAS (0-10) with retrospective duration of at least 6 months
* Low back pain attributed to mechanical as opposed to infectious, neoplastic or inflammatory causes
* Age 18-65
* English speaking
* Male or female
* Mental capacity sufficient to provide informed consent
* Able to commit to up to 27 study meetings over a period of 5 months.

Exclusion Criteria:

* Impairment of hearing, speech, vision, mobility or English fluency sufficient to interfere with participation in the study
* Current or anticipated receipt of payments from Workmen's Compensation or other insurance for disability attributed to low back pain.
* Reports any prior treatment with Structural Integration (Rolf or other varieties, including "structural massage")
* Plans to initiate additional treatment for back pain during the period of the study other than usual rehabilitation care provided at Spaulding Medford clinic, particularly massage or other manual therapy (e.g. chiropractic, osteopathic)
* Unresolved musculoskeletal pathology of the lower limbs
* Pregnancy
* Clinical judgment by Spaulding Medford medical director that the candidate will require either surgery or epidural analgesia within the next five months.
* Alcohol of substance abuse
* Any implanted medical device (e.g. cardio-pacemaker, shunts)
* Prior discectomy or implantation of rods, screws or plates (bulging disc without radicular pain is not exclusionary; hip or shoulder replacement is not exclusionary)
* Current medication with coumadin or prednisone, chronic use of steroid medications, daily use of narcotic analgesics.
* Current diagnosis with any of the following

  1. Balance problems due to vestibular or other neurological impairments
  2. Osteoporosis (osteopenia is not exclusionary)
  3. Fibromyalgia
  4. Severe or progressive neurological deficits, including neuromotor impairment
  5. Any hypercoagulation condition
  6. Eczema, skin infections, deep vein thrombosis
  7. Burns or other acute trauma including unhealed bone fractures or open wounds.
  8. Psychiatric illness not well controlled, or current episode of exacerbated major depressive disorder.
* Any other major medical condition that has not been stabilized, or that would impair the patient's ability to complete the activities required by the study
* Body Mass Index >= 40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Patient rated visual analogue scale (0-10) disturbingness of low back related pain retrospective for one weeks. | 20 weeks

SECONDARY OUTCOMES:
Total score on the Roland Disability Scale | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Jacobson EE, Meleger AL, Bonato P, Wayne PM, Langevin HM, Kaptchuk TJ, Davis RB. Structural integration as an adjunct to outpatient rehabilitation for chronic nonspecific low back pain: a randomized pilot clinical trial. Evid Based Complement Alternat Med. 2015;2015:813418. doi: 10.1155/2015/813418. Epub 2015 Apr 7. PMID 25945112